CLINICAL TRIAL: NCT05666557
Title: Evaluation of the Erector Spinae Muscle Biomechanical Characteristics in Different Position and the Change After Receiving Myofascial Release.
Brief Title: Evaluation of the Erector Spinae Muscle in Different Position and the Change After Receiving Myofascial Release.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMUH110-REC2-071
Record Dates: First submitted 2022-11-09; First posted 2022-12-28 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Low Back Pain
Keywords: Muscle tension tester; muscle characteristics; erector spinae muscles; different postures; myofascial release
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- manual erector spinae myofascial realease (Experimental): Myofascial release is performed by a therapist. The patient prone and using two pillows, one on the head and the other under the abdomen, flexing the lumbar spine maximally under the abdomen with the erector spinae in extension. The therapist will then perform 3 sets of 15 reps with a 1-minute rest between sets with myofascial loosening using standard massage techniques.
  Interventions: Other: manual erector spinae myofascial realease
- self-myofascial release technique (Experimental): Use a roller (roller) to release fascia. The subject stand beside the wall and roll back and forth 15 times as a group, rest for one minute in between, and do a total of 3 groups.
  Interventions: Other: self-myofascial release technique

INTERVENTIONS:
Other: manual erector spinae myofascial realease — The subjects first positioned the third, fourth, and fifth lumbar vertebrae in a relaxed lying position, about 2-3 cm away from the left and right sides (depending on the size of the subjects' muscles). And then in six postures (prone, prone with leg raise, sit straight , slouch sitting, stand straight and slouch standing), MyotonPRO was used to test the above-mentioned 8 points in these position.
  Subjects will undergo a pre-mobilization assessment to see if MyotonPRO can detect changes in the erector spinae muscle properties, including changes in muscle tone, stiffness, and elasticity, under different test positions. After physical therapist manual mobilization, MyotonPRO's erector spinae muscle biomechanical data was collected again for data analysis to determine MyotonPRO could objectively quantify changes in erector spinae biomechanical characteristics.
  Arms: manual erector spinae myofascial realease
Other: self-myofascial release technique — The subjects first positioned the third, fourth, and fifth lumbar vertebrae in a relaxed lying position, about 2-3 cm away from the left and right sides (depending on the size of the subjects' muscles). And then in six postures (prone, prone with leg raise, sit straight , slouch sitting, stand straight and slouch standing), MyotonPRO was used to test the above-mentioned 8 points in these position.
  Subjects will undergo a pre-mobilization assessment to see if MyotonPRO can detect changes in the erector spinae muscle properties, including changes in muscle tone, stiffness, and elasticity, under different test positions. After self mobilization by roller, MyotonPRO's erector spinae muscle biomechanical data was collected again for data analysis to determine MyotonPRO could objectively quantify changes in erector spinae biomechanical characteristics.
  Arms: self-myofascial release technique

SUMMARY:
The purpose of this experiment is to evaluate whether MyotonPRO can quantify the changes in the muscle characteristics of the erector spinae in different postures and after myofascial relaxation, and to test the validity of the muscle tone tester.

DETAILED DESCRIPTION:
In clinical practice, manual muscle testing (MMT) and Modified Ashworth scale (MAS) grading systems are often used to assess muscle tension and tension. Although these methods are considered feasible, because these methods are mainly classified based on the subjective perception of the evaluator, the reliability and accuracy of the evaluation results are often questioned. Therefore, we should seek a way to objectively evaluate muscle tension with biomechanical properties and quantitative data to solve these deviations. MyotonPRO (Myoton AS, Tallinn, Estonia) is a tester that uses biomechanical principles to collect muscle tension status. This handheld muscle tension tester uses mechanical pressure and reaction force feedback to calculate through biomechanical conversion. The tone, stiffness and elasticity of the muscle are expressed as quantitative data. There have been many use reports showing that the muscle tone meter has the feasibility of quantifying muscle tone.

The erector spinae is one of the most important back muscles of the human body. After contraction, the entire spine can be erected, allowing the upper body to stand upright. When the posture changes, such as: sitting posture, hunchback, bending over, erector spinae will be stretched or continuously contracted due to different postures, resulting in changes in muscle characteristics. Therefore, if the erector spinae is used improperly for long-term poor posture, the erector spinae is easily damaged due to heavy burden, which can easily cause back pain. Myofascial release (myofascial release) is a soft tissue massage method that loosens the fascia with hands. By changing the mechanical properties of the muscles, it can loosen over-tension or tense muscles. It is the most commonly used by physical therapists to loosen muscles. One of the operation techniques. However, there is no literature to quantify the effect of myofascial mobilization. The purpose of this experiment is to evaluate whether MyotonPRO can quantify the changes in the muscle characteristics of the erector spinae in different postures and after myofascial relaxation, and to test the validity of the muscle tone tester.

ELIGIBILITY:
Inclusion Criteria:

age 20-65 healthy adult

Exclusion Criteria:

1. Radicular neurological signs
2. spinal deformity e.g.scoliosis, spondylolisthesis
3. infection or tumor
4. Rheumatologic conditions
5. Previous spinal surgery
6. History of hip or pelvic disorder that required treatment
7. male BMI> 27 and female BMI> 26

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-05-11 (Actual); Primary Completion 2021-07-05 (Actual); Study Completion 2022-06-06 (Actual)

PRIMARY OUTCOMES:
Muscle tone of manual erector spinae myofascial release | 10 minutes
  Use MyotonPRO (Myoton AS, Tallinn, Estonia) to assess the muscle tone (Hz)
muscle stiffness of manual erector spinae myofascial realease | 10 minutes
  use MyotonPRO (Myoton AS, Tallinn, Estonia) to assess the muscle stiffness (N/m)
muscle elasticity of manual erector spinae myofascial realease | 10 minutes
  use MyotonPRO (Myoton AS, Tallinn, Estonia) to assess the muscle elasticity (ln(first wave peak/second wave peak))
muscle tone of self-myofascial release technique | 10 minutes
  use MyotonPRO (Myoton AS, Tallinn, Estonia) to assess the muscle tone (Hz)
muscle stiffness of self-myofascial release technique | 10 minutes
  use MyotonPRO (Myoton AS, Tallinn, Estonia) to assess the muscle stiffness (N/m)
muscle elasticity of self-myofascial release technique | 10 minutes
  use MyotonPRO (Myoton AS, Tallinn, Estonia) to assess the muscle elasticity (ln(first wave peak/second wave peak))

CONTACTS AND LOCATIONS:
Overall Officials: Heng-Yi Lin, Bachelor, Principal Investigator — Yueh-Ling Hsieh's bachelor student
Locations (1):
- China Medical University, Taichung, Taiwan

REFERENCES:
- [Background] Aarrestad DD, Williams MD, Fehrer SC, Mikhailenok E, Leonard CT. Intra- and interrater reliabilities of the Myotonometer when assessing the spastic condition of children with cerebral palsy. J Child Neurol. 2004 Nov;19(11):894-901. doi: 10.1177/08830738040190110801. PMID 15658795
- [Background] Jennings AG, Seedhom BB. The measurement of muscle stiffness in anterior cruciate injuries -- an experiment revisited. Clin Biomech (Bristol). 1998 Mar;13(2):138-140. doi: 10.1016/s0268-0033(97)00085-5. PMID 11415781
- [Background] Bizzini M, Mannion AF. Reliability of a new, hand-held device for assessing skeletal muscle stiffness. Clin Biomech (Bristol). 2003 Jun;18(5):459-61. doi: 10.1016/s0268-0033(03)00042-1. PMID 12763442
- [Background] Blackburn JT, Norcross MF, Cannon LN, Zinder SM. Hamstrings stiffness and landing biomechanics linked to anterior cruciate ligament loading. J Athl Train. 2013 Nov-Dec;48(6):764-72. doi: 10.4085/1062-6050-48.4.01. Epub 2013 Jun 14. PMID 24303987
- [Background] Brashear A, Zafonte R, Corcoran M, Galvez-Jimenez N, Gracies JM, Gordon MF, McAfee A, Ruffing K, Thompson B, Williams M, Lee CH, Turkel C. Inter- and intrarater reliability of the Ashworth Scale and the Disability Assessment Scale in patients with upper-limb poststroke spasticity. Arch Phys Med Rehabil. 2002 Oct;83(10):1349-54. doi: 10.1053/apmr.2002.35474. PMID 12370866
- [Background] Brocherie F, Millet GP, Girard O. Neuro-mechanical and metabolic adjustments to the repeated anaerobic sprint test in professional football players. Eur J Appl Physiol. 2015 May;115(5):891-903. doi: 10.1007/s00421-014-3070-z. Epub 2014 Dec 7. PMID 25481506